CLINICAL TRIAL: NCT02551640
Title: Improving Physical Activity Behavior in Patients With High Cardio-metabolic Risk Using a Multi-modal mHealth Intervention: a 2-arm Randomized Controlled Trial
Brief Title: Improving Physical Activity Through a mHealth Intervention in Cardio-metabolic Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015P000765
Record Dates: First submitted 2015-09-10; First posted 2015-09-16 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State; Hypertension; Prehypertension; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Hypertension; Prehypertension; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): * Receive a Samsung smartphone
  * Receive the FeatForward app
  * Receive a Samsung smartwatch
  * Continue to receive medical care as usual
  Interventions: Other: FeatForward App (on study smartphone)
- Group B (No Intervention): * Receive a Samsung smartphone
  * Receive a Samsung smartwatch
  * Continue to receive medical care as usual

INTERVENTIONS:
Other: FeatForward App (on study smartphone) — The FeatForward mobile app will have the following features:
  Messaging: Educational messages tailored to user's medical conditions and motivational messages tailored to user's stage of change.
  Tracking: Ability to track physical activity, weight, blood pressure, blood glucose and heart rate.
  Community: Users in later stages of change able to encourage and motivate one another through groups.
  Educational Library: To provide educational tips and health information. Provider Engagement: Ability for physicians to view patient data, and send messages to patients.
  Monthly depression assessments: The app will prompt users to complete a monthly voluntary depression assessment.
  Social Support: Those using the FeatForward app will also have access to a Facebook group.
  Arms: Group A

SUMMARY:
The goal of this study is to explore the effects of FeatForward on physical activity and cardio-metabolic risk factors. The study will be implemented as a 2-arm randomized controlled trial (RCT) comparing the effects of FeatForward in patients assigned to use the application versus a control group who will not use the app over a 6-month follow-up period. The investigators hypothesize that subjects using FeatForward will be more physically active and will achieve greater improvements in their cardio-metabolic risk (CMR) factors than a usual care control group that will not use the app over a 6-month period.

DETAILED DESCRIPTION:
TextToMove (TTM) was a dynamic text messaging program which the investigators developed in 2012 with the goals of increasing physical activity in patients with type 2 diabetes mellitus (T2DM), improving self-management of the disease, and lowering HbA1c levels. TTM has since been evaluated in a PHRC-approved randomized controlled trial. In our current proposed study, the investigators plan to convert TTM into a mobile application for smartphone use, with increased and improved functionality and with the potential for easy translation to additional use cases. The investigators used feedback gathered from users and observations from the previous trial to shape the development plan for this second iteration, aptly named "FeatForward." The FeatForward app will be hyper-personalized to users and to respond specifically to individual users' behavior patterns so that the application feels like an intelligent health coach partnering with users to achieve better health outcomes. What defines FeatForward from TTM are additional features, including the incorporation of machine learning components for the messaging algorithm, tailoring of message frequency based on users' activity levels, integration of patient data into the electronic medical records through the Remote Monitoring Data Repository, inputs to improve the generalizability of feedback regarding health metrics (e.g., weight, blood glucose), as well as a community feature to enable interactions with other similar patients and a comprehensive educational library.

FeatForward's primary goal is to help users increase their level of physical activity. Physical inactivity has been identified as one of the leading risk factors contributing to the rising rates of chronic diseases. And despite being the most common cardio-metabolic risk (CMR) factor, it also happens to be the easiest to target. Current estimates suggest that over half (52%) of adults in the United States do not meet the recommended physical activity levels. A number of studies to date have demonstrated the dose-response protective effect of increasing physical activity on the development of diabetes and cardiovascular disease. Therefore, the investigators hypothesize that FeatForward will help users to increase their physical activity levels and also lead to improvements in cardio-metabolic risk factors compared to usual care controls that will not use the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of any of the following: pre-diabetes, Type 2 Diabetes Mellitus (T2DM), pre-hypertension, hypertension, and/or obesity (Body Mass Index (BMI) ≥ 30 kg/m2).

  * T2DM: Glycated Hemoglobin (HbA1c) >7.0%
  * Hypertension: Blood Pressure (BP) of 140/90 mmHg
  * Pre-diabetes: HbA1c >5.7% and BMI ≥ 25 kg/m2
  * Pre-hypertension: BP of 130/90 mmHg and family history of high BP
* Willingness to attend all 3 study visits
* Ability to read and speak fluent English
* Physical independence (i.e., ability to walk without assistance)
* Ability to consent for oneself
* Willingness to switch to a provided Samsung smartphone and appropriate phone plan to use as a primary phone for the 6-month study duration
* Willingness to wear a Samsung smartwatch during all hours excluding sleep for the duration of the study

Exclusion Criteria:

* Participants with severe depression assessed by scoring ≥20 on the PHQ-8 screening questionnaire for depression
* Self-reported eating disorder and/or other psychiatric disorders
* Current or recent participation (within 3 months) in a weight loss program
* Prior or planned bariatric surgery procedure
* Use of medications known to cause significant (≥ 5%) long-term changes in body weight or BP
* Pregnancy or plans to get pregnant within 6 months of enrollment
* Disability, dementia or neurological deficits, and other medical or surgical conditions preventing participants from engaging in self-care
* Serious co-morbid conditions (e.g., terminal cancers, end-stage renal disease) that preclude safe participation in moderate levels of physical activity, under discretion of the participants' primary care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Differences in the change in physical activity levels between control and intervention groups as measured by daily physical activity measured by the Gear Fit device provided to participants in both groups | 3 & 6 months

SECONDARY OUTCOMES:
Differences in the change in body weight between control and intervention groups | 3 & 6 months
Differences in the change in HbA1c between control and intervention groups | 3 & 6 months
Differences in the change in fasting blood glucose between control and intervention groups | 3 & 6 months
Differences in the change in blood pressure between control and intervention groups | 3 & 6 months
Differences in the change in waist circumference between control and intervention groups | 3 & 6 months
Differences in the change in serum lipids between control and intervention groups | 3 & 6 months
Differences in the change in C-reactive protein between control and intervention groups | 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Mass General: Charlestown Healthcare Center, Charlestown, Massachusetts
  - Mass General Revere HealthCare Center, Revere, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kohl HW 3rd. Physical activity and cardiovascular disease: evidence for a dose response. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S472-83; discussion S493-4. doi: 10.1097/00005768-200106001-00017. PMID 11427773
- [Background] Kelley DE, Goodpaster BH. Effects of exercise on glucose homeostasis in Type 2 diabetes mellitus. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S495-501; discussion S528-9. doi: 10.1097/00005768-200106001-00020. PMID 11427776
- See also: Centers for Disease Control and Prevention. Chronic Diseases and Health Promotion. 2012 — http://www.cdc.gov/chronicdisease/overview/index.htm.
- See also: Control and Prevention. Physical Activity. — http://www.cdc.gov/physicalactivity/data/facts.html.